CLINICAL TRIAL: NCT05577585
Title: Ketamine Therapy in Obsessive-compulsive Disorder and Its Effects on Neuropsychological Function Under Stress in a Cross-over Trial
Brief Title: Ketamine in OCD: Efficacy and Effects on Stress and Cognition
Acronym: KET-OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christoph Kraus, Ap. Prof. PD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: v6 05.05.2025
Record Dates: First submitted 2022-09-25; First posted 2022-10-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Obsessive-Compulsive Disorder; Psychiatric Disorder
Keywords: Ketamine; stress testing
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Mental Disorders | interventions — Ketamine; Midazolam; Therapeutics

STUDY DESIGN:
Intervention Model Description: This study will apply a randomized, double blind, comparator-controlled cross-over design.
  The order of treatment modality will be randomized and double-blind. Participants will undergo one infusion of ketamine and midazolam as comparator. They will be assigned to one of two sequenced treatment groups, with one group first receiving verum and after 14 days the comparator infusion, the other group vice versa. The randomization into these two sequence groups will be stratified for symptom severity, defined as moderate (YBOCS baseline >16) or severe (YBOCS baseline ≥25). The randomized cross-over phase is followed by an optional open-label continuation with 8 ketamine infusions. Open-label participants are compared to a treatment as usual group.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine (Active Comparator): Participants will undergo one infusion of ketamine as active comparator. (R,S-ketamine 50mg/ml solution for injection, dose: 0,5 mg per kg bodyweight) Both medications will be diluted in 100 ml saline and will be adjusted for infusion over 40 minutes, administered with a syringe pump.
  Interventions: Drug: Ketamine 50 MG/ML Blinded; Drug: Ketamine 50 MG/ML Open Label
- Midazolam (Placebo Comparator): Participants will undergo one infusion of midazolam as comparator. (0,045 mg/kg bodyweight) Both medications will be diluted in 100 ml saline and will be adjusted for infusion over 40 minutes, administered with a syringe pump.
  Interventions: Drug: Midazolam
- Treatment as Usual (Active Comparator): Participants will receive standard-of-care treatment-which may include psychotherapy, pharmacotherapy, physiotherapy, ergotherapy, or a combination of these-at the discretion of the treating physician, independently of the study.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Drug: Ketamine 50 MG/ML Blinded — See also Arm description
  Other Names: Randomized Controlled Phase Intervention 1
  Arms: Ketamine
Drug: Midazolam — See also Arm description
  Other Names: Randomized Controlled Phase Intervention 2
  Arms: Midazolam
Drug: Ketamine 50 MG/ML Open Label — Open Label Follow Up (up to 8 Infusions)
  Other Names: Continuation Phase Intervention 1
  Arms: Ketamine
Other: Treatment as Usual (TAU) — Treatment as Usual may include psychotherapy, pharmacotherapy, physiotherapy, ergotherapy, or a combination of these-at the discretion of the treating physician, independently of the study.
  Other Names: Continuation Phase Intervention 2
  Arms: Treatment as Usual

SUMMARY:
The main goal of this trial is to demonstrate therapeutic efficacy of low dose ketamine in patients with OCD. We expect that ketamine will alleviate symptoms in the hours following application, but also - if effective - that the anti-OCD effects might last for several days after a single infusion.

DETAILED DESCRIPTION:
This study will apply a randomized, double blind, comparator-controlled cross-over design and will be conducted at the Department of Psychiatry and Psychotherapy of the Medical University of Vienna. We will include 30 participants with a primary diagnosis of OCD. Participants will undergo ketamine and comparator infusions in either inpatient- or outpatient settings to assess the therapeutic capabilities of ketamine in OCD. Furthermore, participants' neurocognitive function and stress responses will be tested with four neurocognitive tasks and a cold pressor test paradigm. Also EEG measurements will take place during and before infusions in this phase. Study subjects will be given an option to participate in an open-label follow up with up to 8 infusions over a period of a month. Open-label ketamine treatment will be compared to treatment as usual. After finishing open label treatment an additional EEG measurement will take place.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of obsessive-compulsive disorder
* A score of 16 or higher on the Yale-Brown Obsessive Compulsive Scale and ability to provide written informed consent
* At least one previous treatment for OCD

Exclusion Criteria Experimental Group:

* Any history of current or past psychotic disorder
* A manic episode within the preceding three years
* Current or unstable remitted substance abuse or dependence except nicotine
* Pregnancy or elevated risk of becoming pregnant during study duration (desire to have children) and refusal to utilize a proper method of contraception
* Any current severe personality disorder except comorbid anankastic personality disorder
* Morbus Raynaud
* Inability to follow the study protocol or adhere to operational requirements
* Current and unstable suicidality
* Unstable hypertension
* Untreated hyperthyroidism
* Any unstable cardiovascular disease
* Untreated disorders severely affecting the HPA-axis (M.Addison, M.Cushing)
* Current pharmacological therapy severely affecting the HPA-axis like corticosteroids or ACTH

Exclusion Criteria Treatment as Usual Group:

* Any history of current or past psychotic disorder
* A manic episode within the preceding three years
* Current or unstable remitted substance abuse or dependence except nicotine
* Any current severe personality disorder except comorbid anankastic personality disorder
* Current and unstable suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change of OCD symptoms (Y-BOCS) | In total 7 YBOCS assessments will take place between week 1 and 5.
  There will be a change of severity of obsessive and compulsive symptoms seven days after ketamine infusion compared to midazolam infusion as measured with the Yale-Brown Obsessive Compulsive Scale (Y-BOCS; score range 0-40, with higher scores indicating greater severity).

SECONDARY OUTCOMES:
Change of OCD symptoms (OCD-VAS) | in each arm 24 hours after infusion
  There will be a change in patients' severity of obsessive and compulsive symptoms as measured with the Obsessive-Compulsive Disorder Visual Analog Scale (OCD-VAS; score range 0-600, with higher scores indicating greater severity) 24 hours after ketamine infusion compared to midazolam infusion.
Change of OCD symptoms (Y-BOCS) | in each arm 24 hours after infusion
  There will be a change in patients' severity of obsessive and compulsive symptoms as measured with the Yale-Brown Obsessive Compulsive Scale (Y-BOCS; score range 0-40, with higher scores indicating greater severity) 24 hours after ketamine infusion compared to midazolam infusion.
Change of OCD symptoms (OCD-VAS) | in each arm 1 week after the infusion
  There will be a change of symptoms over the course of seven days after ketamine infusion compared to midazolam infusion as measured with the Obsessive-Compulsive Disorder Visual Analog Scale (OCD-VAS; score range 0-600, with higher scores indicating greater severity) area under the curves.
Change in neuropsychological function | in each arm 24 hours after infusion
  There will be a change in neuropsychological function after 24 hours after ketamine infusion compared to midazolam infusion as measured by four neurocognitive tests (N-Back, WCST, SSRT, ToH)
Change in cortisol response | in each arm 24 hours after infusion
  There will be a change in cortisol response to stress 24 hours after ketamine infusion compared to midazolam infusion.
Change of vegetative stress response (heart rate) | in each arm 24 hours after infusion
  There will be a change of vegetative stress response 24 hours after ketamine infusion compared to midazolam infusion as measured by heart rate.
Change of vegetative stress response (blood pressure) | in each arm 24 hours after infusion
  There will be a change of vegetative stress response 24 hours after ketamine infusion compared to midazolam infusion as measured by blood pressure.
Change of vegetative stress response (stress VAS) | in each arm 24 hours after infusion
  There will be a change of vegetative stress response 24 hours after ketamine infusion compared to midazolam infusion as measured with subjective stress VAS.
Change in OCD symptoms (OCD-VAS) | One month after start of open-label treatment
  Difference of the Obsessive-Compulsive Disorder Visual Analog Scale (OCD-VAS; score range 0-600, with higher scores indicating greater severity) scores a month after open-label treatment compared to treatment as usual, tested in a per protocol set.
Change in OCD symptoms (YBOCS) | One month after start of open-label treatment
  Difference of the Yale-Brown Obsessive Compulsive Scale (Y-BOCS; score range 0-40, with higher scores indicating greater severity) scores a month after open-label treatment compared to treatment as usual, tested in a per protocol set.
Changes in EEG frequency bands | EEG measurements will take place before (5 minutes resting state EEG) and during both infusions of the blinded phase as well as after the open label phase (10 minutes resting state and 5 minutes vigilance EEG).
  There will be distinct changes in EEG frequency bands during ketamine infusion compared to midazolam. EEG will be recorded using a standard 32-channel montage. The following frequency bands will be analyzed at each channel: Delta (0.5-4 Hz), Theta (4-8 Hz), Alpha (8-13 Hz), Beta (13-30 Hz), and Gamma (>30 Hz).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kraus, MD PhD, Principal Investigator — Medical University of Vienna, Department of Psychiatry and Psychotherapy
Locations (1):
- Medical University of Vienna, Department of Psychiatry and Psychotherapy, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No